CLINICAL TRIAL: NCT06705478
Title: An Open-Label, Randomized Controlled Trial of Pramipexole Versus Escitalopram to Treat Major Depressive Disorder (MDD) and Comorbid MDD With Mild Neurocognitive Disorder (MND) in Persons With HIV
Brief Title: Pramipexole Versus Escitalopram to Treat Major Depressive Disorder (MDD) and Comorbid MDD With Mild Neurocognitive Disorder (MND) in Persons With HIV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Cipla Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5402
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder; Mild Neurocognitive Disorder; HIV
Keywords: Comorbid MND
MeSH Terms: conditions — Depressive Disorder, Major; Neurocognitive Disorders | interventions — Escitalopram

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Pramipexole ER (Experimental)
  Interventions: Drug: Pramipexole ER
- Arm 2: Escitalopram (Experimental)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Pramipexole ER — Tablets self-administered orally
  Arms: Arm 1: Pramipexole ER
Drug: Escitalopram — Tablets self-administered orally
  Arms: Arm 2: Escitalopram

SUMMARY:
A phase II, randomized, open-label, two-arm clinical trial evaluating the safety and efficacy of pramipexole extended release (ER) versus escitalopram for the treatment of major depressive disorder (MDD) and comorbid MDD with mild neurocognitive disorder (MND) in persons with HIV (PWH). Participants will be assessed comprehensively and briefly at intercurrent visits to monitor for toxicity, response to therapy, and to assess for dose changes.

An optional sub-study to evaluate treatment impact on the cerebrospinal fluid (CSF) profile will be conducted in a subset of 36 participants.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection.
* Diagnosis of MDD.
* On current ART regimen for at least 90 days prior to study entry with no interruption in treatment greater than 7 consecutive days.
* No plans to change ART while on study.
* Plasma HIV-1 RNA levels of less than 200 copies/mL obtained within 90 days prior to enrollment.
* Study candidates previously treated for depression are eligible provided the study candidate's last dose of antidepressant taken is at least 4 weeks prior to study entry, with the exception of fluoxetine, which the last dose taken must have been at least 8 weeks prior to study entry.
* Laboratory values obtained within 30 days prior to study entry that meet protocol criteria as determined by the site investigator of record.
* Study candidates of child-bearing potential must have a negative serum or urine pregnancy test performed at screening and within 2 days prior to study entry.
* Study candidates of child-bearing potential who are participating in sexual activity that could lead to pregnancy must agree to use at least one highly effective method for contraception.

Exclusion Criteria:

* Active suicidality, and/or severe MDD, psychotic disorders, manic or hypomanic symptoms occurring in the context of bipolar disorder type I or II, or cyclothymic disorder, or another current Axis I diagnosis judged by the investigator to interfere with the trial.
* Study candidate self-report of depressive symptoms that have persisted for over 50 percent of waking hours and for over 50 percent of days over the 24 months prior to study entry.
* Severe, active alcohol or substance use disorder by DSM-5-TR criteria in the 6 months prior to study entry.
* Active alcohol or substance use judged by the investigator to interfere with the trial.
* Any acute infection within 14 days prior to study entry.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 90 days prior to study entry.
* Active coronary artery disease (CAD) or myocardial infarction (MI) within 180 days prior to study entry.
* Presence of rheumatoid arthritis, Sjogren's syndrome, systemic lupus erythematosus (SLE), dermatomyositis, ulcerative colitis, Crohn's disease, or other chronic inflammatory conditions.
* Immune reconstitution inflammatory syndrome (IRIS) or a history of IRIS within 180 days prior to study entry.
* Unstable or advanced liver disease.
* Receipt of medications judged by the site investigator to significantly influence depression or neurocognitive function within 30 days prior to study entry.
* Non-HIV-associated neurological disorder comorbidity.
* Diagnosis of epilepsy with antiepileptic drug treatment.
* Untreated HCV infection and HCV viremia.
* Current CNS malignant tumor or CNS opportunistic infection (OI).
* Current systemic malignant tumor or of a current systemic AIDS-defining OI.
* History of completed treatment of CNS or systemic malignant tumor within the 5 years prior to study entry.
* History of completed treatment of CNS OI within the 5 years prior to study entry.
* Documented history of completed treatment of systemic AIDS-defining OI, as well as Mycobacterium Tuberculosis Infection, within the 180 days prior to study entry.
* New diagnosis of syphilis or treatment for syphilis within the 180 days prior to study entry.
* History of neurosyphilis.
* Severe chronic obstructive pulmonary disease.
* Congestive heart failure (CHF).
* Use of systemic steroids daily (except testosterone).
* Diseases that cause a known bleeding diathesis.
* Immunostimulant therapies and trials of non-FDA-approved ARV medications within 30 days prior to study entry.
* Immunosuppressive medications if judged by the investigator to affect study outcomes.
* Currently pregnant, planning to become pregnant during the study period, or currently breastfeeding.
* Known allergy/sensitivity or any hypersensitivity to the study drugs or their formulations.
* Study candidates on prohibited medications at the time of screening will be excluded from study participation.

Inclusion Criteria for Participants at US Sites Who Consent to the Lumbar Puncture (LP) Procedure:

* Non-focal neurological examination. Study candidates with focal findings should have expert assessment for mass effect prior to the LP.
* Laboratory values that meet LP protocol criteria as determined by the site investigator.
* No history of a positive syphilis testing per local testing algorithms or clinical documentation of prior syphilis treatment.

Exclusion Criteria for Participants at US Sites who Consent to the LP Procedure:

* Current use of anti-coagulants.
* Known presence of intracerebral mass or lesion that is judged to affect the safety of an LP.
* Known presence of an active CNS infection that could alter CNS/CSF inflammatory measures.
* Known allergy to lidocaine.
* Individuals who are unable to safely tolerate an LP due to physical limitation or condition.
* Body mass index (BMI) greater than 40 kg/m^2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory-II (BDI-II/BDI-2) total score defined as the sum of all symptom scores | Baseline, Week 24
Occurrence of Grade ≥3 Adverse Events (AEs) or Grade ≥2 neuropsychiatric AEs related to study treatment | From study treatment administration through Week 24
Occurrence of Grade ≥2 neuropsychiatric AEs related to study treatment | From study treatment administration through Week 24

SECONDARY OUTCOMES:
Change in major depressive disorder (MDD) caseness, defined as the number of symptoms present from 0 to 9, of the symptoms of major depressive disorder | Baseline, Week 24
Complete remission of the major depressive episode defined as a score of 0 on all of the 9 symptoms | Baseline, Week 24
Change in neuropsychological (NP) z-score as assessed through 4 composite domain scores | Baseline, Week 24
  Each domain score is calculated as the average of the z-scores from the tests within the domain:
  * Outcome Domain 1: Cognitive Efficiency (Color Trails 1 and 2)
  * Outcome Domain 2: Verbal Learning and Memory (HVLT-R Learning Trials 1-3 Total and HVLT-R Delayed Recall)
  * Outcome Domain 3: Motor Skills (Grooved Pegboard, Non-dominant hand)
  * Outcome Domain 4: Language (Category Fluency Test [Animals])
Change in the medical outcomes study (MOS)-HIV mental health functioning summary score defined by the MOS-HIV Users Manual | Baseline, Week 24
Change in the MOS-HIV cognitive functioning subscale score defined by the MOS-HIV Users Manual | Baseline, Week 24
Occurrence of Grade ≥3 AEs or Grade ≥2 neuropsychiatric AEs (regardless of judged relationship to study treatment) | From study treatment administration through Week 24
Occurrence of Grade ≥2 neuropsychiatric AEs (regardless of judged relationship to study treatment) | From study treatment administration through Week 24
Number of participants with plasma HIV-1 RNA less than 50 copies/mL | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Karl Goodkin, MD, PhD, Study Chair — Neuropsychiatrist Consultant
Locations (40):
- United States (25):
  - Alabama CRS, Birmingham, Alabama
  - University of California, Los Angeles CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - Harbor University of California, Los Angeles Center CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Whitman-Walker Institute, Inc. CRS, Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS (Site ID 31786), Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Columbia Physicians & Surgeons (P&S) CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Houston Advancing Research Team CRS, Houston, Texas
- Gaborone CRS, Gaborone, Botswana
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra, India
- Kenya (2):
  - Moi University Clinical Research Center (MUCRC) CRS, Eldoret, Rift Valley
  - Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS, Kericho, Rift Valley
- Blantyre CRS, Blantyre, Malawi
- Nutrición-Mexico CRS, Mexico City, Tlalpan, Mexico
- Barranco CRS, Lima, Peru
- De La Salle Medical and Health Sciences Institute - Angelo King Medical Research Center (DLSMHSI-AKMRC), Dasmariñas, Cavite, Philippines
- Durban International CRS, Mount Edgecombe, South Africa
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Pathum Wan, Bangkok
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
- Joint Clinical Research Centre (JCRC)/Kampala CRS, Kampala, Uganda
- Hanoi Medical University (HMU), Hanoi, Vietnam
- Milton Park CRS, Milton Park, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.
URL: https://actgnetwork.org/submit-a-proposal/

REFERENCES:
- [Background] Goodkin K, Evering TH, Anderson AM, Ragin A, Monaco CL, Gavegnano C, Avery RJ, Rourke SB, Cysique LA, Brew BJ. The comorbidity of depression and neurocognitive disorder in persons with HIV infection: call for investigation and treatment. Front Cell Neurosci. 2023 Apr 28;17:1130938. doi: 10.3389/fncel.2023.1130938. eCollection 2023. PMID 37206666
- [Background] Cysique LA, Brew BJ, Bruning J, Byrd D, Costello J, Daken K, Ellis RJ, Fazeli PL, Goodkin K, Gouse H, Heaton RK, Letendre S, Levin J, Aung HL, Mindt MR, Moore D, Mullens AB, de Almeida SM, Munoz-Moreno JA, Power C, Robbins RN, Rule J, Rajasuriar R, Savin MJ, Taylor J, Trunfio M, Vance DE, Wong PL, Woods SP, Wright EJ, Rourke SB. Cognitive criteria in HIV: greater consensus is needed. Nat Rev Neurol. 2024 Feb;20(2):127-128. doi: 10.1038/s41582-024-00927-1. No abstract available. PMID 38228906
- [Background] Goodkin K, Patten SB. Depressive Symptomatology, Syndromal Depression, and HIV-Associated Neurocognitive Disorder (HAND). Can J Psychiatry. 2018 May;63(5):284-286. doi: 10.1177/0706743718754537. No abstract available. PMID 29668329